CLINICAL TRIAL: NCT03190018
Title: A Feasibility Study of Peritoneal Dialysis With CLS PD, Which Removes Toxins and Maintains a Stable Ultrafiltration by Continuously Regenerating a Recirculating Intraperitoneal Fluid, in Patients With End Stage Renal Disease, ESRD, With PD Therapy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Triomed AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Tmed-005 (Gothenburg)
Record Dates: First submitted 2017-05-27; First posted 2017-06-16 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2017-05

CONDITIONS: Peritoneal Dialysis

STUDY DESIGN:
Intervention Model Description: Intervention study, pilot/feasibility for proof of concept of peritoneal dialysis with the Carry Life System for Peritoneal Dialysis (CLS PD)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group with CLS PD device (Experimental): Aim of the intervention is to evaluate the adsorbs of uremic toxins and certain ions with Purcart and the evaluation of the glucose-salt solution ability to achieve stable osmolality. The intervention is during an eight hour study session.
  Interventions: Device: lCarry Life System Peritoneal Dialysis (CLS PD)

INTERVENTIONS:
Device: lCarry Life System Peritoneal Dialysis (CLS PD) — The assigned intervention is with the CLS PD device in patients currently receiving peritoneal dialysis for the duration of one study session. A temporary Pigtail catheter is inserted on the same morning as the study session and removed after the session on the same day.

SUMMARY:
The study is a proof-of-concept of peritoneal dialysis with the Carry Life System for Peritoneal Dialysis (CLS PD). The extra-corporeally absorption of uremic toxins and certain ions from the recirculated peritoneal fluid by the Purcart are evaluated together with the achievement of a stable intraperitoneal osmolarity.

DETAILED DESCRIPTION:
Each patient will be studied during a daytime treatment session of 8 hours. After the inclusion criteria have been met the patient will undergo a Personal Dialysis Capacity test (PDC) to establish the characteristics of the peritoneal membrane, which is required for the individual glucose-salt setting in the device. An ECG and coagulation status will also be performed at this visit.

The clinical study requires the insertion of a temporary catheter (Pigtail) in addition to the patients existing standard PD catheter, and it will be inserted on the morning of the study session. Once the temporary catheter is in situ the peritoneal cavity is filled with a standard glucose based PD solution. Heparin will be added to the PD solution to prevent clogging of the CLS PD. The device is then connected to the catheters and the temporary catheter is used for inflow and positioned in the upper right abdominal quadrant whereas the standard PD catheter in the lower quadrant is used for outflow.

During the study session, a glucose-salt solution will be delivered at a set rate according to individual prescriptions based on the PDC-test and a dosage table based on an algorithm. The osmolarity of the intraperitoneal fluid should be approximately 325 mOsmol/L to obtain an average ultrafiltration of roughly 100 ml/h. It is possible to adjust the delivery rate of the glucose-salt solution during the study session to maintain the desired osmolarity.

The Purcart used for removal of uremic toxins requires replacement after 4 hours of treatment. The use of two Purcarts during the eight-hour study session will provide adequate information with regard to the efficacy of toxin removal.

After the study session, the temporary catheter will be removed and the patient will be hospitalized overnight for observation. The patient will resume their previous PD therapy 36 hours after the study session. The patient's experience of the treatment will be recorded and a follow-up will be performed within 1 week after the study session.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, >18 years of age.
* Prevalent PD patients with ESRD on stable PD without clinical signs of dehydration
* Obtained written consent to participate in the study.
* Negative pregnancy test in females of childbearing age.

Exclusion Criteria:

* Active malignant disease.
* On-going infection.
* HIV and/or hepatitis positive.
* Pregnant, breastfeeding or women of childbearing potential without adequate contraceptive precautions.
* Abdominal hernias.
* Previous major abdominal surgery.
* Any coagulation disorders.
* Anticoagulant therapy within 7 days prior to the study session.
* Allergy to Ecvacillin or Heparin
* Decompensated heart failure
* Conditions except the previous that the Investigator assesses as unsuitable for participation.
* Participation in other clinical trials, which can interfere with this study, within one month before inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
The change in uremic toxins during the study session | During the eight-hour study session
  Measure the uremic toxins before and after the study session to calculate their removal
Maintain stable intraperitoneal osmolarity | During the eight-hour study session
  Measurement of Glucose and Sodium in the intraperitoneal fluid during the study session
Measure ultrafiltered volume | During the eight-hour study session
  The calculated difference between total output minus total fluid intake

SECONDARY OUTCOMES:
Open questions associated with the CLS PD | During eight-hour study session
  The patient will answer open questions objectively describing the portability of the device, sensation associated with the transfer of intraperitoneal fluid in and out of the abdomen and other treatment related viewpoints.
Any Adverse Event (AE) or Serious Adverse Event (SAE) and any Adverse Device Effect (ADE) or Serious Adverse Device Effect (SADE). | Followed during a three week period from visit 2 to visit 4 (1 day follow-up)
  Electrolytes and glucose will be measured both in the blood and the intraperitoneal fluid during the study sessions. The incidence of treatment emergent adverse events or adverse device events occurring during the study

CONTACTS AND LOCATIONS:
Overall Officials: Ola Samuelsson, MD, Principal Investigator — Renal Unit, Sahlgrenska University Hospital, Gothenburg. Sweden
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götalands Regionen, Sweden

IPD SHARING:
Plan to Share IPD: No